CLINICAL TRIAL: NCT01974700
Title: Seizure Prophylaxis in Aneurysm Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment - since the start of the study in 2013, only 17 subjects have consented. Of those, only 8 completed the study.
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCBS-0001
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Intracranial Aneurysms; Seizures
MeSH Terms: conditions — Intracranial Aneurysm; Seizures | interventions — Levetiracetam

ARMS (2):
- Levetiracetam (Active Comparator)
  Interventions: Drug: Levetiracetam
- No anti-epileptic treatment (No Intervention)

INTERVENTIONS:
Drug: Levetiracetam — 500 mg intravenous dose during the operative case then 500 mg orally twice a day for a total of seven days
  Arms: Levetiracetam

SUMMARY:
Seizures are a potential complication of surgical repair of intracranial aneurysms. In order to prevent seizures, many surgeons administer prophylactic anti-epileptic medication during the intra-operative and post-operative period, however, such practice is not supported by clinical data. Retrospective review found the incidence of postoperative seizures was higher in those who received anti-epileptics versus those who did not. The goal is to examine the utility of levetiracetam (Keppra) for seizure prophylaxis in patients undergoing surgical repair of unruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years)
2. Presence of intracranial aneurysm (without rupture)
3. Treating surgeon has recommended surgical repair of the aneurysm.

Exclusion Criteria:

1. History of seizures within last 10 years
2. History of epilepsy
3. History of prior stroke
4. Currently prescribed medication with anti-epileptic activity (keppra,dilantin, tegretol, lamictal, topamax, etc.)
5. Brain tumor
6. Pregnant or nursing woman
7. Known levetiracetam allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 17 were consented, 3 were screen failures, 5 were lost to follow up and one was withdrawn from the study.
Period: Overall Study
Arm/Group | Levetiracetam | No Anti-epileptic Treatment
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | No Anti-epileptic Treatment | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Seizure
Description: Reported via patient in follow-up phone call.
Time Frame: 6 mo - 1 Year from Operative Procedure
Measure: Number; unit: participants
Arm/Group | Levetiracetam | No Anti-epileptic Treatment
Number analyzed (Participants) | 5 | 3
participants | 0 | 1

2. Secondary Outcome: Number of Participants Who Returned to Daily Activities.
Description: The number who had returned to daily activities in the timeframe of 6-12 months, inclusion of those that returned to most of daily activities.
Time Frame: 6 months - 12 months
Measure: Number; unit: participants
Arm/Group | Levetiracetam | No Anti-epileptic Treatment
Number analyzed (Participants) | 5 | 3
participants | 5 | 1

3. Secondary Outcome: Number of Participants Who Returned to Work
Description: The number who had returned to work in the timeframe of 6-12 months, inclusion of those that returned to part-time.
Time Frame: 6 months - 12 months
Measure: Number; unit: participants
Arm/Group | Levetiracetam | No Anti-epileptic Treatment
Number analyzed (Participants) | 5 | 3
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: within 1 year
Arm/Group | Levetiracetam | No Anti-epileptic Treatment
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/3
Other Adverse Events (participants affected / at risk) | 1/5 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=5) | No Anti-epileptic Treatment (N=3)
rehospitalization for seizures (Nervous system disorders) | 0 | 1
benzodiazepine withdrawal rehospitalization (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=5) | No Anti-epileptic Treatment (N=3)
nausea (Gastrointestinal disorders) | 1 | 0
itching (General disorders) | 1 | 0
intraoperative rupture (Injury, poisoning and procedural complications) | 0 | 1
partial seizures (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes